CLINICAL TRIAL: NCT04718727
Title: Olanzapine for the Prevention of Postoperative Nausea and Vomiting After Laparoscopic Surgery in High-risk Patients: A Randomized Controlled Trial
Brief Title: Olanzapine for the Prevention of Postoperative Nausea and Vomiting
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Amani Hassan Abdel-Wahab (Other)
Responsible Party: Sponsor-Investigator, Amani Hassan Abdel-Wahab, assistant professor, Assiut University
Organization: Assiut University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IRB: 17300536
Record Dates: First submitted 2021-01-17; First posted 2021-01-22 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Postoperative Nausea
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Olanzapine

STUDY DESIGN:
Intervention Model Description: All patients will receive oral 10, 5 mg Olanzapine or placebo one hour preoperative
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Placebo Comparator): patients will receive oral placebo tablets one hour preoperatively
  Interventions: Drug: Placebo
- Group 2 (Active Comparator): patients will receive oral 5 mg Olanzapine tablets one hour preoperatively
  Interventions: Drug: 5 mg Olanzapine Tablets
- Group 3 (Active Comparator): patients will receive oral 10 mg Olanzapine tablets one hour preoperatively
  Interventions: Drug: 10 mg Olanzapine Tablets

INTERVENTIONS:
Drug: Placebo — oral Placebo tablets one-hour preoperatively
  Arms: Group 1
Drug: 5 mg Olanzapine Tablets — oral 5 mg Olanzapine tablets one-hour preoperatively
  Other Names: zyprexa
  Arms: Group 2
Drug: 10 mg Olanzapine Tablets — oral 10 mg Olanzapine tablets one-hour preoperatively
  Other Names: zyprexa
  Arms: Group 3

SUMMARY:
Nausea and vomiting (PONV) remain a common problem in surgical units. Even after two or three prophylactic antiemetic interventions, patients with all four of the Apfel risk factors for PONV have an estimated 30 to 40% chance of suffering PONV. Olanzapine as an antiemetic represents a new use of an antipsychotic drug.

DETAILED DESCRIPTION:
Aim of the Research, to compare the effects of oral 10 and 5 mg Olanzapine for the Prevention of Postoperative Nausea and Vomiting

ELIGIBILITY:
Inclusion Criteria:

* ASA I and II patients
* undergoing ambulatory laparoscopic gynecologic surgery with general anesthesia
* patients have at least two of the four Apfel risk factors for PONV2
* Lack of history of psychiatric and psychotic illnesses.

Exclusion Criteria:

* ASA III and ≥ IV patients
* Psychological diseases
* History of chemotherapy
* have a pre-existing vestibular disorder or history of dizziness or preexisting nausea or vomiting in the 24 h before surgery, or were being treated with regular antiemetic therapy including systemic corticosteroids.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 132 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
nausea and/or vomiting score | first 24 hours postoperative
  the occurrence of nausea and/or vomiting by nausea score

CONTACTS AND LOCATIONS:
Overall Officials: Amani H Abdel-wahab, MD, Principal Investigator — Assiut University
Locations (2):
- Egypt (2):
  - Assiut university hospitals, Asyut, Assiut Governorate
  - Assiut university, Asyut

IPD SHARING:
Plan to Share IPD: No